CLINICAL TRIAL: NCT06601725
Title: Clusterin Level Determination and Its Association With Metabolic Syndrome in Patients With Polycystic Ovary Syndrome
Brief Title: Clusterin Level and Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: 2011-KAEK-25 2021/02-06
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Polycystic Ovary Syndrome; Ovulation Disorder
Keywords: clusterin; metabolic syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Biospecimen Retention: Samples Without DNA — Blood samples were collected after at least 12 hours of fasting, 5 mL from the antecubital vein, with the patient in a sitting position using a vacutainer. The samples were placed in a gel tube (biochemistry tube) and centrifuged at 4000 rpm for 5 minutes. Storage conditions were ensured. The samples were stored in a cabinet at -80 degrees Celsius in the genetics laboratory. Clusterin levels were measured using the BT LAB Human Clusterin (CLU) ELISA kit, with min-max values of 0.5-300 ng/ml.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phenotype A: Phenotype A was characterized by metabolic syndrome
  Interventions: Diagnostic Test: Clusterin level
- Phenotype B: phenotype B was characterized by the absence of metabolic syndrome
  Interventions: Diagnostic Test: Clusterin level
- Phenotype C: phenotype C was characterized by hyperandrogenism
  Interventions: Diagnostic Test: Clusterin level
- Phenotype D: phenotype D was characterized by the absence of hyperandrogenism
  Interventions: Diagnostic Test: Clusterin level

INTERVENTIONS:
Diagnostic Test: Clusterin level — Clusterin plays a role in inflammation and oxidative stress processes such as metabolic syndrome, insulin resistance, and atherosclerosis

SUMMARY:
Clusterin, a protein involved in metabolic syndrome, insulin resistance, and metabolic disorders associated with inflammation and oxidative stress such as atherosclerosis, Alzheimer's and some malignancies, has elevated levels in metabolic syndrome, PCOS, and the combination of these two groups. Clusterin could be used as an inflammatory marker to predict PCOS and metabolic syndrome.

DETAILED DESCRIPTION:
The study included 118 women diagnosed with PCOS according to the Rotterdam criteria and 62 age-matched healthy women without cardiovascular risk factors. The patients diagnosed with PCOS were also classified into phenotypes. No interventional examination was requested for patients A, B, C, and D, except for hormonal tests and blood collection for Human Clusterin. The demographic and clinical characteristics of all patients were compared, with the primary outcome being blood Clusterin levels. The secondary outcomes are blood Clusterin levels in women with and without metabolic syndrome in addition to PCOS, the relationship between PCOS phenotypes and Clusterin levels, and the relationship between Clusterin levels and clinical and laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 45,
* natural bilateral ovaries and no functional cysts on transvaginal ultrasound.

Exclusion Criteria:

* who have hyperandrogenism/hyperandrogenemia
* who have non-classical congenital adrenal hyperplasia (17 OHP value >2 nmol/L)
* who have thyroid disease (TSH >5 mlU/L),
* women with hyperprolactinemia (Prolactin>30 mlU/mL)
* patients taking hormonal drugs or ovulation induction agents.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 118 women who were diagnosed with polycystic ovary syndrome (PCOS) according to the Rotterdam criteria, as well as 62 healthy women of the same age without any cardiovascular risk factors. Patients diagnosed with PCOS were classified into four phenotypes: A, B, C, and D. Phenotype A was characterized by metabolic syndrome, phenotype B was characterized by the absence of metabolic syndrome, phenotype C was characterized by hyperandrogenism, and phenotype D was characterized by the absence of hyperandrogenism.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
CLusterin level | 7 months
  primary outcome is the measurement of blood Clusterin (Apolipoprotein J) levels in healthy women with and without PCOS

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı Yenigül, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No